CLINICAL TRIAL: NCT07154966
Title: Prospective Evaluation of Chemotherapy-Induced Taste Alterations, Sarcopenia, and Malnutrition in Patients With Gynecologic Malignancies Treated With Carboplatin and Paclitaxel
Brief Title: Taste Alteration, Sarcopenia, and Malnutrition in Gynecologic Cancer Patients Receiving Carboplatin-Paclitaxel Chemotherapy
Acronym: GYM-TASTE
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncologist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK-2025-122; AEŞH-EK-2025-122 (Other: Ankara Etlik City Hospital Clinical Research Ethics Committee)
Record Dates: First submitted 2025-08-24; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Ovarian Cancer (OvCa); Fallopian Tube Cancers; Endometrial Cancer; Chemotherapy-Induced Taste Alteration; Cancer-Associated Malnutrition; Cancer-Associated Sarcopeni
Keywords: Gynecologic malignancies; Ovarian cancer; Fallopian tube cancer; Endometrial cancer; Chemotherapy; Taste alteration (dysgeusia); Malnutrition; Sarcopenia; PG-SGA; CITAS; Supportive oncology
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Dysgeusia; Malnutrition; Sarcopenia | interventions — CP protocol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carboplatin-Paclitaxel Cohort: Patients with histologically confirmed non-metastatic ovarian, fallopian tube, or endometrial cancer receiving six cycles of standard carboplatin-paclitaxel chemotherapy (carboplatin AUC 5 + paclitaxel 175-200 mg/m² every 21 days). Assessments at baseline (before chemotherapy), after Cycle 3 (~9 weeks), and after Cycle 6 (~18 weeks). Evaluations: CITAS, PG-SGA, CT-based SMI, ECOG performance status, laboratory parameters, anthropometrics.
  Interventions: Other: Standard Chemotherapy (Carboplatin-Paclitaxel)

INTERVENTIONS:
Other: Standard Chemotherapy (Carboplatin-Paclitaxel) — Standard-of-care chemotherapy with carboplatin (AUC 5, every 21 days) and paclitaxel (175-200 mg/m², every 21 days) for six cycles. No additional drugs, dose modifications, or alternative regimens introduced.

SUMMARY:
This observational study aims to evaluate chemotherapy-induced taste alterations, sarcopenia, and malnutrition in patients with gynecologic malignancies (ovarian, fallopian tube, and endometrial cancer) treated with standard carboplatin and paclitaxel. Eligible patients will receive six cycles of chemotherapy (carboplatin area under the curve [AUC] 5 + paclitaxel 175-200 mg/m², every 21 days), and assessments will be performed at baseline (before chemotherapy), after the 3rd cycle (~9 weeks), and after the 6th cycle (~18 weeks). Validated tools will be used, including the Chemotherapy-Induced Taste Alteration Scale (CITAS, Turkish validated, range 18-90; higher scores indicate greater severity of dysgeusia), the Patient-Generated Subjective Global Assessment (PG-SGA, Turkish validated, range 0-35; higher scores indicate worse nutritional status), and Computed Tomography (CT)-based Skeletal Muscle Index (SMI) at the L3 vertebra level.

DETAILED DESCRIPTION:
Gynecologic malignancies, including ovarian, fallopian tube, and endometrial cancers, are among the leading causes of morbidity and mortality in women. Standard first-line treatment with carboplatin and paclitaxel improves survival but can cause adverse effects such as dysgeusia (taste alteration), weight loss, sarcopenia, and malnutrition. Chemotherapy-induced dysgeusia may reduce oral intake, alter dietary preferences, and worsen protein-energy malnutrition, accelerating muscle loss and functional decline. Sarcopenia and myosteatosis, assessed using CT-based SMI measurements at the L3 vertebra, have been shown to affect chemotherapy tolerance and prognosis.

This single-center observational study at Ankara Etlik City Hospital enrolled 102 female patients with non-metastatic ovarian, fallopian tube, or endometrial cancer undergoing six cycles of carboplatin-paclitaxel. Systematic evaluations included CITAS, PG-SGA, CT-based SMI, Eastern Cooperative Oncology Group (ECOG) performance status (range 0-5; higher scores indicate worse functional status), laboratory parameters, and anthropometric measures.

Primary objectives:

Incidence and severity of chemotherapy-induced taste alterations

Changes in nutritional status (PG-SGA)

Changes in skeletal muscle index (SMI)

Secondary objectives:

Correlation between CITAS and PG-SGA scores with dietary intake and chemotherapy adherence

Correlation between sarcopenia/malnutrition and chemotherapy-related toxicities (hematologic toxicities, fatigue)

Changes in ECOG performance status and functional capacity

Exploratory: correlations with inflammatory markers (C-reactive protein [CRP], albumin)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-metastatic ovarian, fallopian tube, or endometrial cancer
* Planned to receive adjuvant or neoadjuvant carboplatin-paclitaxel regimen (carboplatin AUC 5 + paclitaxel 175-200 mg/m² every 21 days)
* No prior chemotherapy
* Age ≥ 18 years, female
* Completion of 6 cycles of carboplatin-paclitaxel treatment
* Availability of CT imaging at baseline, after third cycle, and after sixth cycle
* Ability to provide written informed consent

Exclusion Criteria:

* Metastatic disease or palliative treatment setting
* Treatment with regimens other than carboplatin-paclitaxel or weekly protocols
* Prior systemic therapy (e.g., immunotherapy, targeted therapy) Initial treatment discontinuation due to progression, toxicity, or patient preference
* Missing CT imaging at required timepoints
* Pregnancy or breastfeeding
* Cognitive impairment or inability to provide informed consent
* Severe comorbid conditions (e.g., uncontrolled cardiac disease, end-stage renal failure, advanced liver failure)
* Inability to comply with study assessments or follow-up visits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult female patients (≥18 years) with histologically confirmed non-metastatic ovarian, fallopian tube, or endometrial cancer who are receiving adjuvant or neoadjuvant carboplatin-paclitaxel chemotherapy at Ankara Etlik City Hospital. A total of 102 patients will be enrolled. Participants must have completed six cycles of standard chemotherapy and have available CT imaging at baseline, after the third cycle, and after the sixth cycle to allow prospective evaluation of taste alterations, nutritional status, and sarcopenia.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of chemotherapy-induced taste alterations | Baseline (before chemotherapy), at the end of Cycle 3 (each cycle is 21 days, ~9 weeks), and at the end of Cycle 6 (each cycle is 21 days, ~18 weeks).
  Chemotherapy-Induced Taste Alteration Scale (CITAS, Turkish validated). Range: 18-90; higher scores = greater severity of dysgeusia. Cut-offs: 18-30 = minimal, 31-60 = moderate, 61-90 = severe.
Change in skeletal muscle index (SMI) at L3 vertebra level | Baseline (before chemotherapy), at the end of Cycle 3 (each cycle is 21 days, ~9 weeks), and at the end of Cycle 6 (each cycle is 21 days, ~18 weeks).
  CT-based skeletal muscle area at L3, normalized for height (cm²/m²). Cut-offs: Female <38.5 cm²/m², Male <52.4 cm²/m² define sarcopenia.
Change in nutritional status measured by PG-SGA | Baseline (before chemotherapy), at the end of Cycle 3 (each cycle is 21 days, ~9 weeks), and at the end of Cycle 6 (each cycle is 21 days, ~18 weeks).
  Patient-Generated Subjective Global Assessment (PG-SGA, Turkish validated). Range: 0-35; higher = worse nutritional status. Cut-offs: 0-1 = no intervention, 2-3 = education, ≥4 = intervention, ≥9 = intensive support.

SECONDARY OUTCOMES:
Impact of taste alterations on nutritional intake and treatment adherence | Baseline (before chemotherapy), at the end of Cycle 3 (each cycle is 21 days, ~9 weeks), and at the end of Cycle 6 (each cycle is 21 days, ~18 weeks).
  Correlation between CITAS scores (18-90; higher = worse dysgeusia) and PG-SGA scores (0-35; higher = worse nutritional status) with appetite changes, dietary preferences, and completion of planned chemotherapy cycles.
Association between sarcopenia/malnutrition and chemotherapy-related toxicities | Throughout chemotherapy (baseline to end of Cycle 6, each cycle is 21 days, ~18 weeks).
  Correlation of CT-based SMI (Female <38.5, Male <52.4) and PG-SGA (0-35) with toxicities: neutropenia, anemia, thrombocytopenia, fatigue.
Change in ECOG performance status and functional capacity | Baseline (before chemotherapy), at the end of Cycle 3 (each cycle is 21 days, ~9 weeks), and at the end of Cycle 6 (each cycle is 21 days, ~18 weeks).
  Eastern Cooperative Oncology Group (ECOG) performance status. Range: 0-5; higher = worse performance. Cut-offs: 0 = fully active, 1 = restricted, 2 = ambulatory, 3 = limited self-care, 4 = disabled, 5 = death.

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Ankara Etlik City Hospital Medical Oncology Department; Osman Sütcüoğlu, MD, Principal Investigator — Gazi University Medical Oncology Department, Ankara; Ömür Berna Öksüzoğlu, MD, Principal Investigator — Ankara Etlik City Hospital Medical Oncology Department
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No